CLINICAL TRIAL: NCT03387527
Title: Using Decision Analysis to Enhance Decision-Making Regarding Prostate Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE7817
Record Dates: First submitted 2017-12-22; First posted 2018-01-02 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Prostate Cancer
Keywords: Decision Aid
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prostate Cancer Decision Aid (Experimental): The research intervention will be exposure to the screening decision aid. Patients will receive standardized counseling including population based risks and benefits of prostate cancer screening. Then, patients will be given opportunity to review the screening decision aid prior to offering a decision on whether or not to undergo prostate cancer screening. The patient decision aid will be a computer application that generates predicted risks associated with prostate cancer.
  Interventions: Behavioral: Prostate cancer decision aid

INTERVENTIONS:
Behavioral: Prostate cancer decision aid — Patients will undergo standardized counseling and individualized counseling with the screening decision aid. The screening decision aid is a computer program that provides individual patients estimates of their risks of prostate cancer diagnosis, prostate cancer related death, or death from any cause
  Other Names: screening decision aid

SUMMARY:
The purpose of this study is to evaluate a new counseling tool for patients deciding whether or not to undergo prostate cancer screening. This screening decision aid is a computer program that provides individual patients estimates of their risks of prostate cancer diagnosis, prostate cancer related death, or death from any cause. The researchers are evaluating whether or not patients find this screening decision aid helpful. As part of this study, participants will be asked for their response on questionnaires.

If patients find the screening decision aid helpful, the researchers will make it available at other clinic locations.

DETAILED DESCRIPTION:
To conduct a feasibility study on implementing the computer-based screening decision aid for prostate cancer screening in a primary care setting during a 60-minute interview. To aid in informed decision making, the screening decision aid will include a graphical representation of predicted probabilities of prostate cancer diagnosis, prostate cancer-specific mortality, death from competing causes based on a man's unique demographic information. The study team will provide standardized counseling followed by individualized counseling with the screening decision aid. It will assess the quality of the decision making process (patient feels knowledgeable, informed of the risks/benefits, feels clear about their values, is involved in the decision), and quality of the decision.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy > 10 years
* Ability to read English

Exclusion Criteria:

* Personal history of prostate cancer
* Personal history of prostate biopsy or prostate surgery
* Prior prostate specific antigen screening in the past year leading up to their scheduled clinic visit
* Cognitive impairment

Ages: 55 Years to 69 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-10-03 (Actual); Study Completion 2018-11-03 (Actual)

PRIMARY OUTCOMES:
Number of initial interviews completed in 60 minutes | 60 minutes from beginning of interview
  To be considered feasible in a busy clinical setting, researchers anticipate 80% of the initial interviews to be completed within the allotted 60-minute interview time.

SECONDARY OUTCOMES:
Health Literacy | 1 month after clinical visit
  Five item scale measuring attitudes towards screening
Patient decisional control preferences | 1 month after clinical visit
  4 item scale where lower scores indicate more positive outcomes from screening
Decisional conflict Scale | 1 month after clinical visit
  16 item scale ranging in a score from 0-4 where higher scores indicate more disagreement
Multidimensional measure of informed choice | 1 month after clinical visit
  10 item true/false scale
Decisional regret scale | 1 month after clinical visit
  5 item questionnaire using 5 point Likert scales where higher scores indicate more disagreement

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Brooks, MD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States